CLINICAL TRIAL: NCT04170595
Title: A Randomized, Multicenter, Phase I/IIa Clinical Study to Evaluate the Tolerability, Safety, Efficacy, Pharmacokinetics and Immunogenicity of GB221 for Injection for the Treatment of HER2-positive Breast Cancer Patients
Brief Title: Clinical Study of Recombinant Anti-HER2 Humanized Monoclonal Antibody for Injection
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Genor Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GENOR GB221-002
Record Dates: First submitted 2019-11-12; First posted 2019-11-20 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: HER2-positive Breast Cancer
MeSH Terms: interventions — Trastuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- GB221,2mg/kg (Experimental): Coprelotamab Injection, 2 mg/kg, Single dose,
  Interventions: Biological: GB221,2 mg/kg
- GB221,6mg/kg (Experimental): Coprelotamab Injection, 6 mg/kg, Single dose,
  Interventions: Biological: GB221,6 mg/kg
- Herceptin,6mg/kg (Active Comparator): Trastuzumab Injection, 6 mg/kg, Single dose,
  Interventions: Biological: Herceptin,6 mg/kg
- GB221,8mg/kg (Experimental): Coprelotamab Injection, 8 mg/kg, Single dose,
  Interventions: Biological: GB221,8mg/kg
- GB221+ Capecitabine (Experimental): Multiple dose groups
  Interventions: Biological: GB221:2mg/kg and Capecitabi:1000mg/kg
- Herceptin+Capecitabine (Active Comparator): Multiple dose groups
  Interventions: Biological: Herceptin:2mg/kg and Capecitabin:1000mg/kg

INTERVENTIONS:
Biological: GB221,2 mg/kg — Single dose, 2mg/kg group: lyophilized powder of Coprelotamab Injection; strength 110mg/bottle; 2 mg/kg for one dose, intravenous infusion, completed for over 90 minutes
  Other Names: Coprelotamab Injection
  Arms: GB221,2mg/kg
Biological: GB221,6 mg/kg — Single dose 6mg/kg group: lyophilized powder of Coprelotamab Injection; strength 110mg/bottle; 6 mg/kg for one dose, intravenous infusion, completed for over 90 minutes
  Other Names: Coprelotamab Injection
  Arms: GB221,6mg/kg
Biological: Herceptin,6 mg/kg — Single dose group: lyophilized powder of Trastuzumab Injection; strength 440 mg/bottle; 6 mg/kg for one dose, intravenous infusion, completed for over 90 minutes
  Other Names: Trastuzumab Injection
  Arms: Herceptin,6mg/kg
Biological: GB221,8mg/kg — Single dose 8mg/kg group: lyophilized powder of Coprelotamab Injection; strength 110mg/bottle; 8mg/kg for one dose, intravenous infusion, completed for over 90 minutes
  Other Names: Coprelotamab Injection
  Arms: GB221,8mg/kg
Biological: GB221:2mg/kg and Capecitabi:1000mg/kg — GB221:Lyophilized powder of Coprelotamab Injection; strength 110mg/bottle; 2mg/kg, the first infusion is completed over 90 minutes. If no serious adverse reaction is observed, the subsequent infusion can be completed over 30 minutes. The administration shall be continued until disease progression or intolerable toxic reactions or ICF withdrawal of subjects. Multiple dose group; Capecitabine:1000mg/kg, orally twice daily (one dose each in the morning and evening; total daily dose of 2000 mg/m2), administration for 2 weeks followed by a 1-week rest period, as a 3-week cycle.
  Arms: GB221+ Capecitabine
Biological: Herceptin:2mg/kg and Capecitabin:1000mg/kg — Herceptin:Lyophilized powder of Trastuzumab Injection; strength 440 mg/bottle; 2mg/kg, the first infusion is completed over 90 minutes. If no serious adverse reaction is observed, the subsequent infusion can be completed over 30 minutes. The administration shall be continued until disease progression or intolerable toxic reactions or ICF withdrawal of subjects. Multiple dose groups; Capecitabine:1000mg/kg, orally twice daily (one dose each in the morning and evening; total daily dose of 2000 mg/m2), administration for 2 weeks followed by a 1-week rest period, as a 3-week cycle.
  Arms: Herceptin+Capecitabine

SUMMARY:
A randomized, multicenter, Phase I/IIa clinical study to evaluate the tolerability, safety, efficacy, pharmacokinetics and immunogenicity after single/multiple administration of recombinant anti-HER2 humanized monoclonal antibody for injection for the treatment of HER2-positive breast cancer patients.

ELIGIBILITY:
For single dose:

Inclusion Criteria:

1. Aged 18 to 65 years;
2. Histopathologically confirmed breast cancer;
3. HER-2 positive (definition: the immunohistochemistry (IHC) test of pathological samples showed HER-2 +++ or immunohistochemistry (IHC) test showed HER-2 ++ and positive FISH amplification test);
4. HER2-positive breast cancer patients who have no lesion after surgery and never received anti-HER-2 treatment;
5. The investigators consider that the subject has recovered from the toxic reactions caused by the previous chemotherapy 4 weeks after the last chemotherapy.
6. The expected survival is 3 months or longer;
7. ECOG performance status is 0, 1 or 2;
8. The left ventricular ejection fraction (LVEF)≥50%;
9. The major organ function is normal and laboratory tests meet relevant criteria:

   l Hematology test:
   * Hb≥90 g/L (no blood transfusion within 14 days);
   * ANC≥1.5×109 /L;
   * PLT≥100×109 /L; l Hepatic and renal function tests:
   * TBIL≤1.5×ULN (upper limit of normal);
   * ALT and AST≤2.5×ULN;
   * Serum Cr ≤ULN;
10. Normal coagulation function test;
11. Voluntarily sign the written informed consent form

Exclusion Criteria:

1. Pregnant or breastfeeding females; or women of childbearing potential who have positive urine pregnancy test; or any subjects who are able to bear or father a child but cannot or are unwilling to adopt medically acceptable effective contraceptive methods during the study period and within 3 months after the end of the study;
2. Subjects who have any of the following cardiac conditions:

   * Unstable angina pectoris;
   * Medical history of congestive heart failure;
   * Previous medical history of myocardial infarction, coronary artery bypass grafting or coronary stent implantation;
   * Clinically significant pericardial diseases and valvular heart diseases;
   * Serious uncontrolled arrhythmia;
   * Any other cardiac diseases which may cause safety risks for patients if they are enrolled in this study;
3. Uncontrolled hypertension (defined as screening systolic blood pressure ≥ 180mmHg and/or diastolic blood pressure ≥110mmHg);
4. Known HIV, HBV or HCV infection;
5. Allergic constitution; known allergic to the components of the investigational product;
6. Have drug abuse history or alcohol addiction history;
7. Participated in other clinical studies within 4 weeks before the initiation of the study;
8. Have complicated diseases which may interfere with study participation or evaluation at the discretion of the investigator, e.g., uncontrolled infection, coagulation disorders and other diseases, or the investigators consider that participation in this study may lead to greater risks for patients.

For multiple dose groups:

Inclusion Criteria:

1. Aged 18 to 65 years;
2. Histopathologically confirmed breast cancer;
3. HER-2 positive (definition: the immunohistochemistry (IHC) test of pathological samples showed HER-2 +++ or immunohistochemistry (IHC) test showed HER-2 ++ and positive FISH amplification test);
4. Patients with metastatic breast cancer who failed to respond to previous chemotherapy and no more than three lines, and never received anti-HER-2 treatment(subjects in single dose group who experienced disease progression but meet other inclusion/exclusion criteria can be enrolled);
5. There is at least one measurable target lesion (based on RECIST 1.1 criteria):

   * According to Response Evaluation Criteria in Solid Tumors (RECIST V1.1), the target lesions must be accurately measured in at least one dimension (refer to appendix 5);
   * No radiotherapy for target lesions;
6. The investigators consider that the subject has recovered from the toxic reactions caused by the previous chemotherapy 4 weeks after the last chemotherapy (subjects who are receiving Xeloda monotherapy and achieve efficacy or stable disease can be enrolled in this study).
7. The expected survival is 3 months or longer;
8. ECOG performance status is 0, 1 or 2;
9. The left ventricular ejection fraction (LVEF)≥50%;
10. The major organ function is normal and laboratory tests meet relevant criteria:

    l Hematology test:
    * Hb≥90 g/L (no blood transfusion within 14 days);
    * ANC≥1.5×109 /L;
    * PLT≥100×109 /L; l Hepatic and renal function tests:
    * TBIL≤1.5×ULN (upper limit of normal);
    * ALT and AST≤2.5×ULN; if there is any hepatic metastasis, ALT and AST ≤5×ULN;
    * Serum Cr ≤ULN;
11. Normal coagulation function test;
12. Voluntarily sign the written informed consent form.

Exclusion Criteria:

1. Pregnant or breastfeeding females; or women of childbearing potential who have positive urine pregnancy test; or any subjects who are able to bear or father a child but cannot or are unwilling to adopt medically acceptable effective contraceptive methods during the study period and within 3 months after the end of the study;
2. Subjects with known or suspected brain metastasis: Subjects with evidence indicating signs or symptoms of brain metastasis are not allowed to participate in this study unless such brain metastasis is excluded by CT or MRI. However, subjects whose brain metastasis lesions have been controlled can be enrolled (no progression within at least 4 weeks after radiotherapy and/or no neurological symptom or sign after surgical resection, treatment with dexamethasone or mannitol is not necessary);
3. Subjects who had disease progression after previous chemotherapy with Xeloda.
4. Subjects who have any of the following cardiac conditions:

   * Unstable angina pectoris;
   * Medical history of congestive heart failure;
   * Previous medical history of myocardial infarction, coronary artery bypass grafting or coronary stent implantation;
   * Clinically significant pericardial diseases and valvular heart diseases;
   * Serious uncontrolled arrhythmia;
   * Any other cardiac diseases which may cause safety risks for patients if they are enrolled in this study;
5. Uncontrolled hypertension (defined as screening systolic blood pressure ≥ 180mmHg and/or diastolic blood pressure ≥110mmHg);
6. Known HIV, HBV or HCV infection;
7. Allergic constitution; known allergic to the components of the investigational product;
8. Have drug abuse history or alcohol addiction history;
9. Participated in other clinical studies within 4 weeks before the initiation of the study;
10. Have complicated diseases which may interfere with study participation or evaluation at the discretion of the investigator, e.g., uncontrolled infection, coagulation disorders and other diseases, or the investigators consider that participation in this study may lead to greater risks for patients.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2014-03-28 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
maximum tolerated dose,MTD | Up to 5 weeks
  To evaluate the efficacy and safety of GB221.
C max | Up to 5 weeks
  C max
AUC (0- t) | Up to 5 weeks
  AUC (0- t)
AUC (0- ∞ ) | Up to 5 weeks
  AUC (0- ∞ )
T max | Up to 5 weeks
  T max
T 1/2 | Up to 5 weeks
  T 1/2
CL/F | Up to 5 weeks
  CL/F
V/F | Up to 5 weeks
  V/F
K e | Up to 5 weeks
  K e

SECONDARY OUTCOMES:
Antidrug antibody, ADA | Up to 5 weeks
  Antidrug antibody, ADA

CONTACTS AND LOCATIONS:
Overall Officials: Ze Fei Jiang, Ph.D, Principal Investigator — Affiliated Hospital of Academy of Military Medical Sciences
Locations (1):
- Affiliated Hospital of Academy of Military Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No